CLINICAL TRIAL: NCT02379182
Title: Randomized Controlled Trial To Evaluate The Effect Of Vitalstim In Patients With Chronic Post-stroke Oropharyngeal Dysphagia
Brief Title: Effect Of Vitalstim In Patients With Chronic Post-stroke Oropharyngeal Dysphagia
Acronym: VITAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pere Clave (Other)
Collaborators: Hospital de Granollers (Other)
Responsible Party: Sponsor-Investigator, Pere Clave, MD, PhD, Hospital de Mataró
Organization: Hospital de Mataró (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VITAL
Record Dates: First submitted 2015-02-27; First posted 2015-03-04 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Deglutition Disorders; Stroke
Keywords: dysphagia; VitalStim; electrical stimulation
MeSH Terms: conditions — Deglutition Disorders; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- Control group (Active Comparator): Will not receive any treatment procedure. Patients allocated in the control group will be treated according to the standard clinical care of patients with dysphagia at our center, that includes: adaptation of fluids, diet and oral hygiene recommendations, and postural and swallowing maneuvers training if necessary.
  Interventions: Behavioral: standard clinical care
- Sensory Group (Experimental): Patients allocated in the sensory group will be treated with transcutaneous electrical stimulation at sensory level. In addition, they will receive the standard clinical care described in the control group. The treatment procedure will consist of the application, at rest, of 80 Hz of transcutaneous electrical stimulus (biphasic, 700 µs) using VitalStim device (Chattanooga Group, Hixson, TN, USA), 2 sessions of 1 hour per day the first week, and 1 hour per day the next week. Sessions will be applied for two weeks. Treatment intensity will be set to 75% of motor threshold and electrode placement, thyro-hyoid (placement 3a described in the VitalStim Certification Program). The motor threshold will be determined by triplicate, as the intensity level at which the patient reports a grabbing or pulling sensation and confirmed by the clinician. Every 10 min, the patient will be asked if the initial sensation is maintained and, if necessary, treatment intensity will be re-adjusted.
  Interventions: Behavioral: standard clinical care; Device: transcutaneous electrical stimulation at sensory level
- Motor Group (Experimental): Patients allocated in the motor group will be treated with transcutaneous electrical stimulation at motor level. In addition, they will receive the standard clinical care of patients with dysphagia described in the control group. The treatment procedure will consist of the application, at rest, of 80 Hz of transcutaneous electrical stimulus (biphasic, 700 µs) using VitalStim device (Chattanooga Group, Hixson, TN, USA), 2 sessions of 1 hour per day the first week, and 1 hour per day the next week. Sessions will be applied from Monday to Friday for two weeks. Treatment intensity will be set to the motor threshold and electrode placement, supra-hyoid. The motor threshold will be determined by triplicate, as the intensity level at which the patient reports a grabbing or pulling sensation and confirmed by the clinician. Every 10 min, the patient will be asked if the initial sensation is maintained and, if necessary, treatment intensity will be re-adjusted.
  Interventions: Behavioral: standard clinical care; Device: transcutaneous electrical stimulation at motor level

INTERVENTIONS:
Behavioral: standard clinical care — adaptation of fluids, diet and oral hygiene recommendations, and postural and swallowing maneuvers training if necessary
Device: transcutaneous electrical stimulation at sensory level — The treatment procedure will consist of the application, at rest, of 80 Hz of transcutaneous electrical stimulus (biphasic, 700 µs) using VitalStim device (Chattanooga Group, Hixson, TN, USA), 2 sessions of 1 hour per day the first week, and 1 hour per day the next week. Sessions will be applied from Monday to Friday for two weeks. Treatment intensity will be set to 75% of motor threshold and electrode placement, thyro-hyoid (placement 3a described in the VitalStim Certification Program). The motor threshold will be determined by triplicate, as the intensity level at which the patient reports a grabbing or pulling sensation and confirmed by the clinician. Every 10 min, the patient will be asked if the initial sensation is maintained and, if necessary, treatment intensity will be re-adjusted.
  Arms: Sensory Group
Device: transcutaneous electrical stimulation at motor level — The treatment procedure will consist of the application, at rest, of 80 Hz of transcutaneous electrical stimulus (biphasic, 700 µs) using VitalStim device (Chattanooga Group, Hixson, TN, USA), 2 sessions of 1 hour per day the first week, and 1 hour per day the next week. Sessions will be applied from Monday to Friday for two weeks. Treatment intensity will be set to the motor threshold and electrode placement, supra-hyoid. The motor threshold will be determined by triplicate, as the intensity level at which the patient reports a grabbing or pulling sensation and confirmed by the clinician. Every 10 min, the patient will be asked if the initial sensation is maintained and, if necessary, treatment intensity will be re-adjusted.
  Arms: Motor Group

SUMMARY:
Prospective, randomized, controlled, three-arm, open-label, blinded analysis. Patients admitted with stroke diagnosis and with suspected dysphagia that meet the initial inclusion and exclusion criteria will be consented into the clinical investigation. Patients who meet the second set of inclusion criteria (dysphagia confirmed by VFS) will be randomized to either active (motor or sensory) or standard treatment (control group) arms.

Subjects included in this clinical investigation will be evaluated at screening, 1-week, 3-months and at 12-months post treatment.

The main aim of the study will be to assess the effect of VitalStim therapy on improving the safety of swallow according to the VFS, after the treatment and at 1-year follow up, on patients with chronic post-stroke OD.

ELIGIBILITY:
Inclusion Criteria:

* Subject is over 18 years of age.
* Subject is suspected of having oropharyngeal dysphagia.
* Subject is able to comply with videofluoroscopy protocol.
* Subject diagnosed with stroke.
* Subject has no previous history of dysphagia.
* Subjects who are able to give voluntary, written informed consent to participate in the clinical investigation and from whom consent has been obtained/ or a consultee has consented on the subjects behalf in line with nationally agreed guidelines concerning adults unable to consent for themselves.
* Subject is not currently participating in any other interventional clinical study.
* Subject is able to comply with the protocol requirements
* Subject scores 0 or 1 on question 1a of NIHSS

Randomization Inclusion Criteria:

• Subject has confirmed dysphagia (PAS of 2 or more on VFS screening or pharyngeal residue).

Exclusion Criteria:

* Subject stroke event occurred less than 3 months ago.
* Subject is pregnant or a nursing mother.
* Subject, in the opinion of the investigator, has advanced dementia
* Subject fitted with a pacemaker or implantable cardiac defibrillator
* Subject is dysphagic from conditions other than stroke
* Subject has been diagnosed with a progressive neurological disorder, such as Parkinson's disease or Multiple Sclerosis.
* Subject with active neoplasm or infection process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-10; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change in Penetration-Aspiration scores | baseline and Post-treatment visit (5 days)
Change in Penetration-Aspiration scores | baseline and 1 year

SECONDARY OUTCOMES:
Incidence of all adverse events | 1 year
Change in pharyngeal residue prevalence | Post-treatment visit (5 days)
Change in pharyngeal residue prevalence | 1 year
Change in EAT-10 scores | Post-treatment visit (5 days)
Change in EAT-10 scores | 1 year
Frequency of chest infections | 1 year
Time from randomisation to death | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Mataró, Mataró, Barcelona, Spain